## Informed Consent Form:

## "Treatment of ulcers associated with hammer, mallet and claw toe deformities in the diabetic patient setting"

## **Declaration from research participant:**

I have received sufficient written and oral information regarding aim, method, advantages and risks to agree to participation in this project

I am conscious that participation is voluntary, and that I can always retract my consent, without giving up my current or future rights in relation to treatment.

I hereby consent to participation in this research project and have been offered a copy of the consent form and the written information regarding this project.

| Research participants name: | |
|---|---|
| Patient ID Number | : |
| Date: | Signature: |
| | elated information regarding, you is discovered during the course of the project you you do <b>not</b> wish to be informed, please mark with x here: |
| Do you wish to be to your treatment: | informed on results of the project after conclusion of the project, and how it pertains |
| Yes No | ) |
| Declaration from | investigator who supplied information: |
| I hereby declare th | at participant has received written and oral information pertaining to the project. |
| To the best of my participation in the | knowledge the given information is sufficient for participant to make decision regarding project. |
| Name of the invest | igator that has given the information: |
| Date: | Signature: |

Version 1.2 01/10-2019 Page 1